CLINICAL TRIAL: NCT04549194
Title: Contribution of L-Tyrosine to Recovery From Operational Strain on Return From External Operation
Acronym: USOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2019PBMD06; 2020-A01658-31 (Other: IDRCB)
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Stress, Psychological
Keywords: L-tyrosine
MeSH Terms: conditions — Stress, Psychological | interventions — Blood Specimen Collection; Tyrosine; Photoplethysmography

STUDY DESIGN:
Intervention Model Description: The study is composed of 2 groups, each of which is composed of 2 arms:
  * External Operation group
    * L-Tyrosine arm
    * Placebo arm
  * Rear Base group
    * L-Tyrosine arm
    * Placebo arm
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The pharmacist, carrying out the packaging and labelling of the treatment units, will ensure the blinding. Neither the participant nor the investigator will know what treatment is being administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tyrosine - External Operation (Experimental): 1-month L-Tyrosine treatment following 4-month external operation
  Interventions: Biological: Blood collection; Drug: L-Tyrosine 500 Mg; Behavioral: Psychological questionnaires; Device: Photoplethysmography
- Placebo - External Operation (Experimental): 1-month Placebo treatment following 4-month external operation
  Interventions: Biological: Blood collection; Behavioral: Psychological questionnaires; Device: Photoplethysmography; Drug: Placebo
- Tyrosine - Rear Base (Experimental): 1-month L-Tyrosine treatment following 4 months at rear base
  Interventions: Biological: Blood collection; Drug: L-Tyrosine 500 Mg; Behavioral: Psychological questionnaires; Device: Photoplethysmography
- Placebo - Rear Base (Experimental): 1-month Placebo treatment following 4 months at rear base
  Interventions: Biological: Blood collection; Behavioral: Psychological questionnaires; Device: Photoplethysmography; Drug: Placebo

INTERVENTIONS:
Biological: Blood collection — A blood sample will be collected before during and after the treatment.
Drug: L-Tyrosine 500 Mg — The participants will be administered 4 capsules of L-Tyrosine 500 mg per oral route daily over 1 month.
  Arms: Tyrosine - External Operation; Tyrosine - Rear Base
Behavioral: Psychological questionnaires — The participants will fill in several psychological questionnaires before, during and after treatment administration:
  * Life Event Checklist
  * Moral injury
  * Posttraumatic Checklist
  * Burnout Assessment Tool
  * State-Trait Anger Expression Inventory-2
  * Ruminative Response Scale - Reconsidered
  * Deployment Risk and Resilience Inventory-2
  * Questionnaire about tobacco use
Device: Photoplethysmography — Photoplethysmography recording will be performed before during and after the treatment.
Drug: Placebo — The participants will be administered 4 capsules of Lactose 500 mg (placebo) per oral route daily over 1 month.
  Arms: Placebo - External Operation; Placebo - Rear Base

SUMMARY:
Operational conditions amplify soldier's constraints and stress factors, upsetting individual and collective adaptive landmarks. The soldier's resistance is strained by the high intensity of stressors, by the long duration of exposure and by their cumulative effect.

This may lead to a state of "operational strain" that refers to chronic stress and the allostatic load imposed by operational constraint.

The investigators believe that operational strain could manifest itself by a kind of accelerated aging of the organism due to the increased allostatic load without sufficient resource restoration (neurotransmitter precursors, partial and repeated sleep deprivation, etc.).

This aging mechanism would be reversible after a sufficient period of resource restoration (sleep, physical activity, adapted diet, etc.).

ELIGIBILITY:
Inclusion Criteria:

* From 18 to 65 years of age

Exclusion Criteria:

* Tyrosine intake within the previous 15 days
* History of neurological or psychiatric disorder
* History of nephrological or endocrine disorder or liver failure
* Hereditary tyrosinemia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Difference between the change in Burnout Assessment Tool (BAT) score following 1-month treatment in each arm | After 1-month treatment
  The Burnout Assessment Tool (BAT) is used to assess burn-out risk. The score ranges from 1 to 5, with higher scores indicating a higher risk of burn-out.

SECONDARY OUTCOMES:
Difference between the change in catecholamine level following 1-month treatment in each arm | After 1-month treatment
  Catecholamine level will be measured in blood before during and after 1-month treatment.
Difference between the change in aminoacid level following 1-month treatment in each arm | After 1-month treatment
  Aminoacid level will be measured in blood before during and after 1-month treatment.
Difference between the change in zonulin level following 1-month treatment in each arm | After 1-month treatment
  Zonulin level will be measured in blood before during and after 1-month treatment.
Difference between the change in Brain-Derived Neurotrophic Factor (BDNF) level following 1-month treatment in each arm | After 1-month treatment
  BDNF level will be measured in blood before during and after 1-month treatment.
Difference between the change in gamma-aminobutyric acid (GABA) level following 1-month treatment in each arm | After 1-month treatment
  GABA level will be measured in blood before during and after 1-month treatment.
Difference between the change in Tumor Necrosis Factor Alpha (TNFα) level following 1-month treatment in each arm | After 1-month treatment
  TNFα level will be measured in blood before during and after 1-month treatment.
Difference between the change in Interleukin-6 (IL6) level following 1-month treatment in each arm | After 1-month treatment
  IL6 level will be measured in blood before during and after 1-month treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recherche Biomédicale des Armées, Brétigny-sur-Orge, France

IPD SHARING:
Plan to Share IPD: Undecided